CLINICAL TRIAL: NCT06545357
Title: Evaluating the Effectiveness of Treating Shoulder Subluxation After Stroke With Modified Acupuncture of Biceps Brachii Muscle, Supraspinatus Muscle and Deltoid Muscles: a Randomized, Double-blind, Controlled Clinical Trial
Brief Title: Effective Treatment of Shoulder Subluxation After Stroke With Modified Acupuncture of Biceps Brachii Muscle, Supraspinatus Muscle and Deltoid Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Collaborators: My-Suong Thi Phan (Unknown); Dieu-Thuong Thi Trinh (Unknown)
Responsible Party: Principal Investigator, Bui Pham Minh Man, medicine doctor, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 702/HDDD-DHYD
Record Dates: First submitted 2024-06-21; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Shoulder Subluxation After Stroke
Keywords: Shoulder subluxation after stroke; Modified acupuncture
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Active Comparator): 36 participants received upright shoulder X-rays before intervention to evaluate shoulder subluxation. Participants of the intervention group were received modified acupuncture to improve the biceps brachii muscle, supraspinatus muscle and deltoid muscle; The degree of shoulder subluxation will be evaluated by X-ray of the shoulder joint after 4 weeks of intervention.
  Interventions: Procedure: Acupuncture
- The control group (Sham Comparator): 36 participants received upright shoulder X-rays before intervention to evaluate shoulder subluxation. Participants of the control group were received conventional electroacupuncture according to The Stomach Channel -Yangming; The degree of shoulder subluxation will be evaluated by X-ray of the shoulder joint after 4 weeks of intervention.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — To conduct this intervention, we used disposable acupuncture needles with the size of 0.30 x 25 mm to acupuncture at biceps brachii muscle, supraspinatus muscle and deltoid muscles or acupoints on The Yang Ming Channel for 20 minutes, frequency ≤ 20 Hz, intensity from 2- 10mA

SUMMARY:
Stroke is the most common emergency in neurology and is also the leading cause of disability, so recovery of movement after stroke is very important. However, a common complication of stroke is shoulder subluxation, which hinders recovery of movement, thereby leading to shoulder pain and increasing the level of disability after stroke. Neuromuscular electrical stimulation affecting the biceps brachii muscle, supraspinatus muscle and deltoid muscles has been proven to be relatively effective in treating shoulder subluxation after stroke. However, this method does not go through the skin, so it is difficult to have a deep impact on the muscles and difficult to cause selective muscle contractions, so the treatment of this disease is still limited. In traditional medicine, modified acupuncture has a mechanism of action similar to neuromuscular electrical stimulation and is a method that passes through the skin, stimulating muscles effectively and selectively. In our study, we wanted to evaluate the effectiveness of treating shoulder subluxation after stroke with modified acupuncture of biceps brachii muscle, supraspinatus muscle and deltoid muscles

DETAILED DESCRIPTION:
Participants and methods: A randomized controlled clinical trial was conducted by comparing the change in shoulder subluxation in post-stroke patients. A total of 72 participants were randomly assigned to 2 groups using GraphPad software on the computer, and the allocation ratio was 1:1. Participants in the intervention group were received modified acupuncture of biceps brachii muscle, supraspinatus muscle and deltoid muscles, while the control group were received conventional electroacupuncture of acupuncture points along The Stomach Channel -Yangming in the shoulder region. The result are the change in the degree of shoulder subluxation according to the qualitative method of Van Langenberghe and Hogan and the quantitative method of Hall J. This study was conducted randomized, controlled and double-blind.

ELIGIBILITY:
Inclusion Criteria:

Patients satisfy all of the following criteria:

* Age enough 18 years old or older.
* Diagnosed with stroke (based on hospital discharge papers or brain CT-scan or brain MRI results, if available).
* During the recovery period (24 hours - 6 months) according to the classification of KNGF 2014.
* Has subluxated shoulder joint (assessed on X-ray of straight shoulder joint according to Van Langenberghe and Hogan criteria)
* Volunteer to sign the consent form to participate in the study.

Exclusion Criteria:

Patients not be selected for the study if they have any one of the following conditions:

* Have previous shoulder pathology not related to stroke such as tumor, infection, scapular instability, winged scapula, brachial plexus injury, periarthritis humeroscapularis (recorded through asking about the patient's history)
* Have skin infections and ulcers in the paralyzed shoulder area.
* Have a blood clotting disorder or lack of clotting factors (recorded through asking the patient's history).
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
The grade of shoulder subluxation was measured according to the qualitative method of Van Langenberghe and Hogan | After 4 weeks of intervention
The grade of shoulder subluxation was measured according to Hall J's quantitative method | After 4 weeks of intervention
Classification of treatment response according to shoulder subluxation grade (the qualitative method of Van Langenberghe and Hogan) | After 4 weeks of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Traditional medicine - University of Medicine and Pharmacy of Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Demographic characteristic and outcome data will be shared
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Result] Wang RY, Chan RC, Tsai MW. Functional electrical stimulation on chronic and acute hemiplegic shoulder subluxation. Am J Phys Med Rehabil. 2000 Jul-Aug;79(4):385-90; quiz 391-4. doi: 10.1097/00002060-200007000-00011. PMID 10892625
- [Result] Koyuncu E, Nakipoglu-Yuzer GF, Dogan A, Ozgirgin N. The effectiveness of functional electrical stimulation for the treatment of shoulder subluxation and shoulder pain in hemiplegic patients: A randomized controlled trial. Disabil Rehabil. 2010;32(7):560-6. doi: 10.3109/09638280903183811. PMID 20136474
- [Result] Manigandan JB, Ganesh GS, Pattnaik M, Mohanty P. Effect of electrical stimulation to long head of biceps in reducing gleno humeral subluxation after stroke. NeuroRehabilitation. 2014;34(2):245-52. doi: 10.3233/NRE-131041. PMID 24419017
- [Result] Van Langenberghe HV, Hogan BM. Degree of pain and grade of subluxation in the painful hemiplegic shoulder. Scand J Rehabil Med. 1988;20(4):161-6. PMID 3232046
- [Result] Hall J, Dudgeon B, Guthrie M. Validity of clinical measures of shoulder subluxation in adults with poststroke hemiplegia. Am J Occup Ther. 1995 Jun;49(6):526-33. doi: 10.5014/ajot.49.6.526. PMID 7645665
- [Result] Pyace Phyo Nyein, Myat Bhone Aung, Thein Than Win, Khin Win Sein. Effects of electrical stimulation to long head of biceps in glenohumeral subluxation after stroke.ResearchGate. 2020;doi:10.13140/RG.2.2.28053.06886